CLINICAL TRIAL: NCT01746303
Title: Omega-3 and Blueberry Supplementation in Age-Related Cognitive Decline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Robert Krikorian, Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R01AG034617-01 (NIH)
Record Dates: First submitted 2012-12-05; First posted 2012-12-10 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Age-related Memory Disorders; Mood Disorders
Keywords: Working memory; Long-term memory; Neurocognition; Dietary supplementation; dementia
MeSH Terms: conditions — Memory Disorders; Mood Disorders; Dementia | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Omega 3 and Blueberry powder (Experimental): This group will receive omega-3 fatty acid and blueberry powder supplement for 24 weeks (6 months)
  Interventions: Dietary Supplement: Omega-3 fatty acid; Dietary Supplement: Blueberry powder
- Omega-3 and placebo powder (Experimental): This group will receive omega-3 fatty acid and placebo powder for 24 weeks (6 months)
  Interventions: Dietary Supplement: Omega-3 fatty acid; Other: Placebo powder
- Placebo oil and blueberry powder (Experimental): This group will receive placebo oil and blueberry powder for 24 weeks (6 months).
  Interventions: Dietary Supplement: Blueberry powder; Other: Placebo oil
- Placebo oil and placebo powder (Placebo Comparator): This group will receive placebo oil and placebo powder for 24 weeks (6 months)
  Interventions: Other: Placebo oil; Other: Placebo powder

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acid — A fixed dose of 2.4 g/day (EPA: 1.6 g, DHA: 0.8 g; 4 capsules/d).
  Other Names: OmegaRx capsules
  Arms: Omega 3 and Blueberry powder; Omega-3 and placebo powder
Dietary Supplement: Blueberry powder — Whole, freeze-dried blueberry powder made of 50%:50% mixture of Tifblue and Rubel blueberries.
  Arms: Omega 3 and Blueberry powder; Placebo oil and blueberry powder
Other: Placebo oil — Corn oil capsules that are identical in size, shape, and color to omega-3 capsules.
  Arms: Placebo oil and blueberry powder; Placebo oil and placebo powder
Other: Placebo powder — Placebo powder matched for color, taste, and sugar content as closely as possible and milled similarly to the blueberry powder.
  Arms: Omega-3 and placebo powder; Placebo oil and placebo powder

SUMMARY:
The aim of this study is to determine the efficacy of 6 months' dietary supplementation with omega-3 fatty acids and whole freeze dried blueberry powder in improving cognition in older adults. The effects of each of these interventions alone will also be assessed in order to determine whether the combined treatment confers synergistic or additive benefit relative to the effect of each therapy.

DETAILED DESCRIPTION:
After meeting inclusion criteria, one hundred-forty men and women, aged 62 to 80 years old, will be enrolled and randomly assigned to one of four groups: 1) omega-3 fatty acid and blueberry powder supplement, 2) omega-3 fatty acid and placebo powder, 3) placebo oil and blueberry powder supplement, or 4) placebo oil and placebo powder. They will participate in a 24-week intervention with major assessments including neuropsychological and functional evaluation at pre-treatment baseline and during the final week of the intervention. In addition, an interim evaluation of neurocognitive function will be conducted at 12 weeks. Subjects will be asked to maintain diet diaries for three periods during the study. Mood will be assessed as a potential covariate of the neurobehavioral outcome measures and data on red blood cell fatty acid content, metabolic parameters, inflammation, and anthropometric factors will be gathered to assess compliance and explore individual differences in response to the intervention and to evaluate potential mechanisms of action.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged 62 to 80 years and older
* age-associated decline operationalized as Clinical Dementia Rating = 0, Auditory Verbal Learning Test cumulative acquisition score between 1.0 standard deviation below and 1.0 standard deviation above the age-corrected mean or Montreal Cognitive Assessment score greater than 25, and Geriatric Depression Scale score less than 16
* ability to comprehend and comply with the research protocol
* provision of written informed consent.

Exclusion Criteria:

* established dementia or neurological disorder including but not limited to probable Alzheimer's Disease, Parkinson's Disease, Frontotemporal dementia, multi-infarct dementia, and leukoencephalopathy
* current or past severe psychiatric disorder such as psychosis or major mood disorder requiring hospitalization and/or causing a change in level of occupational or social functioning
* current or past alcohol or drug abuse disorder causing physiological dependence or change in functional capability (nicotine dependence is permitted)
* diagnosis of diabetes or other metabolic disorder or kidney or liver disease
* use of medication that might affect outcome measures or interact with omega 3 fatty acid supplements such as benzodiazepines, aspirin, and serotonin reuptake inhibitors
* hematological coagulation disorder
* allergy to shellfish or seafood; 8) current supplementation with fish oil or consumption of fish more than once per week.

Ages: 62 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2010-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Working Memory and Executive Ability | 6 months
  The following tests will be administered to measure working memory function:
  * Porteus Maze Test
  * Verbal Primary Memory with Interference Test
  * Letter Number Sequencing Task
  * Controlled Oral Word Production Task

SECONDARY OUTCOMES:
Mood Assessment | 6 months
  The following scale will be used to assess mood:
  * Geriatric Depression Scale
  * Geriatric Anxiety Inventory
Daily Functioning Assessment | 6 months
  The following scale will be used to measure daily functioning:
  - Older Americans Resources and Services Functional Assessment Questionnaire
Long-term memory function | 6 months
  The following assessments will be conducted to measure Long-term memory function:
  * California Verbal Learning Test, Second Edition
  * Visual Nonverbal Recognition Memory Test
  * Verbal Paired Associate Learning Task
  * Spatial Paired Associate Learning Task

OTHER OUTCOMES:
Ancillary Measures | 6 months
  The following measures will be collected:
  * Red blood cell fatty acid composition
  * Inflammatory and metabolic parameters
  * Waist Circumference, Hip Circumference, Height, Body Weight, Blood pressure, Heart rate
  * Urinary anthocyanin studies
  * Diet Diaries

CONTACTS AND LOCATIONS:
Overall Officials: Robert Krikorian, PhD, Principal Investigator — University of Cincinnati; Robert McNamara, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] McNamara RK, Kalt W, Shidler MD, McDonald J, Summer SS, Stein AL, Stover AN, Krikorian R. Cognitive response to fish oil, blueberry, and combined supplementation in older adults with subjective cognitive impairment. Neurobiol Aging. 2018 Apr;64:147-156. doi: 10.1016/j.neurobiolaging.2017.12.003. Epub 2017 Dec 12. PMID 29458842
- [Derived] Boespflug EL, McNamara RK, Eliassen JC, Schidler MD, Krikorian R. Fish Oil Supplementation Increases Event-Related Posterior Cingulate Activation in Older Adults with Subjective Memory Impairment. J Nutr Health Aging. 2016 Feb;20(2):161-9. doi: 10.1007/s12603-015-0609-6. PMID 26812512